CLINICAL TRIAL: NCT02426489
Title: Improving Diagnosis of Breast Cancer by Using a Combined MRI and Positron Emission Mammography (MRI-PEM) System
Acronym: MRI-PEM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Subcontract PI left institution.
Sponsor: Weinberg Medical Physics LLC (Industry)
Collaborators: University of California, Irvine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: WMP-2
Record Dates: First submitted 2015-04-09; First posted 2015-04-27 (Estimated); Last update posted 2021-10-07 (Actual); Status verified 2021-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diagnostic accuracy with MRI alone (No Intervention): The MRI of the breast lesion will be examined. Measures of performance accuracy will be evaluated, including diagnostic sensitivity (true positives divided by true positives and false negatives), diagnostic specificity (true negatives divided by true negatives and false positives), and diagnostic accuracy, defined as the number of correct assessments divided by the number of all assessments.
- Diagnostic accuracy with MRI + PEM image (Experimental): The combined PEM/MRI image will be examined.
  Interventions: Device: MRI + PEM image

INTERVENTIONS:
Device: MRI + PEM image — Effect of positron emission mammography on diagnostic accuracy
  Other Names: flurodeoxyglucose
  Arms: Diagnostic accuracy with MRI + PEM image

SUMMARY:
The purpose of the study is to assess whether the addition of positron emission mammography will add diagnostic value to magnetic resonance imaging of the breast, in patients with lesions of the breast that are suspicious enough to warrant biopsy, or which have been confirmed as containing cancer cells.

DETAILED DESCRIPTION:
70 eligible subjects will be asked to undergo contrast-enhanced MRI studies of the breast containing the lesion. Subjects will be asked to fast for 6 hours prior to the imaging session. Each subject will be tested for glucose, and if the glucose is not too high, the subject will be injected with a dose of radioactive sugar (fluoro-deoxyglucose) which has been shown in other studies to accumulate in breast cancers. The subject will be asked to sit quietly for 30 minutes and to empty the bladder. The subject will then be asked to be re-examined in the MRI scanner with MRI contrast injection. The examination bed will be moved out of the MRI scanner and detectors of the radioactive sugar will be placed near the breast in order to obtain a positron emission mammogram for a 10-minute period. The subject will then leave the MRI suite.

ELIGIBILITY:
Inclusion Criteria:

* Female over 21 years of age;
* with a suspicious lesion found in the breast and recommended for biopsy or have a confirmed diagnosis of cancer;
* and in good health (other than having breast lesions);
* and can lie still in a prone position for 30 minutes in an MRI scanner.

Exclusion Criteria:

* Pregnancy;
* unwilling to give informed consent;
* have implanted prosthetic heart valve,
* pacemaker,
* neurostimulator,
* surgical clips or other metallic implants;
* have engaged in occupations or received orthodontic work which may have caused lodging of ferromagnetic materials in the body;
* are claustrophobic;
* have been allergic to contrast agents;
* are diabetic;
* or have a history of kidney disease.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2016-05-08 (Actual); Study Completion 2016-05-08 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of combination MRI/positron emission mammography (diagnostic accuracy, defined as the number of correct assessments divided by the number of all assessments) | up to 2 years
  Patients with benign disease on biopsy may be followed for up to 2 years after imaging

CONTACTS AND LOCATIONS:
Overall Officials: Irving Weinberg, MD PhD, Principal Investigator — Weinberg Medical Physics LLC

IPD SHARING:
Plan to Share IPD: No